CLINICAL TRIAL: NCT03756090
Title: A Randomized Study Evaluating the Safety and Effects of the Combination of Palbociclib With Epirubicin and Cyclophosphamide Followed by Paclitaxel as Neoadjuvant Therapy in Triple Negative Breast Cancer
Brief Title: The Combination of Palbociclib With ddEC-P as Neoadjuvant Therapy in Triple Negative Breast Cancer
Acronym: PECP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PECP
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer; Breast Diseases; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — palbociclib; Epirubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Arm I: Palbociclib combined with Dose-Dense neoadjuvant chemotherapy for total 16 weeks.
  Interventions: Drug: Palbociclib; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel
- Control group (Placebo Comparator): Arm II: Placebo combined with Dose-Dense neoadjuvant chemotherapy for total 16 weeks.
  Interventions: Drug: Placebo oral capsule; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be administered orally as 125mg capsules, daily on a schedule of 3 weeks (21 days) on, 1 week (7 days) off of a 4 week [28 days] cycle.
  Arms: Experimental group
Drug: Placebo oral capsule — Placebo oral capsule will be administered orally as 125mg capsules, daily on a schedule of 3 weeks (21 days) on, 1 week (7 days) off of a 4 week [28 days] cycle.
  Arms: Control group
Drug: Epirubicin — Epirubicin (90mg/m2, D1) cycled every 14 days for the first 4 cycles.
Drug: Cyclophosphamide — Cyclophosphamide (600mg/m2, D1) cycled every 14 days for the first 4 cycles.
Drug: Paclitaxel — Paclitaxel (80mg/m2, D1) cycled every 14 days for the later 4 cycles.

SUMMARY:
This study will look at effects the combination of palbociclib and dose-dense neoadjuvant chemotherapy may have on triple negative breast cancer tumours which have not yet been treated.

DETAILED DESCRIPTION:
Patients will be randomized to one of two treatment arms (1:1 ratio). Dose-Dense neoadjuvant chemotherapy in the first 8 weeks of will be: epirubicin (90mg/m2) and cyclophosphamide (600mg/m2), followed by paclitaxel (80mg / m2) after 8 weeks, cycled every 14 days for total 8 cycles.

Palbociclib will be administered orally as 125mg capsules, daily on a schedule of 3 weeks (21 days) on, 1 week (7 days) off of a 4 week [28 days] cycle.

Arm I: Palbociclib combined with Dose-Dense neoadjuvant chemotherapy for total 16 weeks.

Arm II: Placebo combined with Dose-Dense neoadjuvant chemotherapy for total 16 weeks.

Note:

Following completion of study therapy, surgery will be scheduled for 18-20 weeks post-randomization.

Post-surgical treatment will be at the discretion of treating clinician, following postoperative pathology.

After week 16 (end of study therapy) all patients should continue Palbociclib for one year.

Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).

ELIGIBILITY:
Inclusion Criteria:

1. female patients, 18 years ≤ age ≤ 80 years；
2. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
3. Histologically confirmed invasive breast cancer（early stage or locally advanced）
4. HER2 negative (HER2+/- by IHC or FISH-)
5. Hormone receptor (ER and PR) negative
6. Cardiovascular: Baseline left ventricular ejection fraction (LVEF)≥55% measured by ECHO
7. Signed informed consent form (ICF)

Exclusion Criteria:

1. Metastatic disease (Stage IV) or inflammatory breast cancer
2. Previous or current history of malignant neoplasms, except for curatively treated: Basal and squamous cell carcinoma of the skin, Carcinoma in situ of the cervix.
3. Clinically relevant cardiovascular disease: Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110);
4. Unable or unwilling to swallow capsules.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
pCR | Through study completion, an average of 1 year.
  Percentage of Participants With Pathological Complete Response (pCR) at the Time of Surgery.

SECONDARY OUTCOMES:
DFS | Following surgery until Year 3
  Disease-free Survival
ORR | Through study completion, an average of 1 year.
  Objective Response Rate (ORR) during neoadjuvant period
AEs | baseline and weekly through 12 months after randomization
  Number and severity of adverse events.Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Ding Xiaowen, DR., Principal Investigator — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: Undecided